CLINICAL TRIAL: NCT03571607
Title: A PHASE 3, MULTICENTER, SINGLE-ARM, OPEN-LABEL STUDY TO ASSESS THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF A SINGLE DOSE OF 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN JAPANESE SUBJECTS AGED 6 TO 64 YEARS WHO ARE CONSIDERED TO BE AT INCREASED RISK OF PNEUMOCOCCAL DISEASE AND WHO ARE NAIVE TO PNEUMOCOCCAL VACCINES
Brief Title: A Safety And Immunogenicity Study Of A 13-valent Pneumococcal Conjugate Vaccine In Japanese Subjects Aged 6 To 64 Years.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1851172; 2018-003054-24 (EudraCT Number)
Record Dates: First submitted 2018-06-20; First posted 2018-06-27 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 13-valent pneumococcal conjugate vaccine (Experimental)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — A single dose (0.5 mL) will be administered intramuscularly into the deltoid muscle at visit 1.
  Other Names: 13vPnC

SUMMARY:
This study is to evaluate the safety, tolerability and immunogenicity of a single dose of 13-valent pneumococcal conjugate vaccine in Japanese subjects aged 6 to 64 years who are considered to be at increased risk of pneumococcal disease and who are naive to pneumococcal vaccines.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males and females aged 6 to <65 years at enrollment.
* Subjects with an increased risk of pneumococcal disease determined by documented medical history, physical examination, and clinical judgment of the investigator.

Exclusion Criteria:

* Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt during study participation.
* End-stage disease including but not limited to metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, or end-stage renal disease with or without dialysis.
* Graft-versus-host disease (GVHD), history of solid organ transplant within 6 months before investigational product administration or history of HSCT, or potential for solid organ transplant or HSCT during study participation.
* Receipt of cytotoxic chemotherapy or blood products within 3 months before investigational product administration or anti-B-cell antibodies within 6 months before investigational product administration through completion of study participation.
* Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components.
* Documented S pneumoniae infection within the past 5 years before investigational product administration.

Ages: 6 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 206 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Japan (8):
  - Daido Clinic, Nagoya, Aichi-ken
  - Nippon Kokan Fukuyama Hospital, Fukuyama, Hiroshima
  - Fukuyama City Hospital, Fukuyama, Hiroshima
  - Kawasaki Municipal Hospital, Kawasaki, Kanagawa
  - Nagano Prefectural Shinshu Medical Center, Suzaka, Nagano
  - Medical Co.LTA PS Clinic, Fukuoka
  - Fukuoka Children's Hospital, Fukuoka
  - National Hospital Organization Kumamoto Medical Center, Kumamoto

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Yamazaki Y, Ikeda M, Imada T, Furuno K, Mizukami T, de Solom R, Shoji Y, Oe M, Aizawa M, Giardina PC, Schmoele-Thoma B, Scott DA. A phase 3, multicenter, single-arm, open-label study to assess the safety, tolerability, and immunogenicity of a single dose of 13-valent pneumococcal conjugate vaccine in Japanese participants aged 6-64 years who are considered to be at increased risk of pneumococcal disease and who are naive to pneumococcal vaccines. Vaccine. 2021 Oct 15;39(43):6414-6421. doi: 10.1016/j.vaccine.2021.08.106. Epub 2021 Sep 23. PMID 34563397
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1851172

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: 6 to <18 Years: Participants aged between 6 to less than (<) 18 years received a single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly on Day 1.
- 13vPnC: 18 to <65 Years: Participants aged between 18 to <65 years received a single 0.5 mL dose of 13vPnC intramuscularly on Day 1.
Period: Overall Study
Arm/Group | 13vPnC: 6 to <18 Years | 13vPnC: 18 to <65 Years
Started | 53 | 153
Vaccinated | 53 | 153
Completed | 53 | 153
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received 1 dose of study vaccine.
Groups:
- 13vPnC: 6 to <18 Years: Participants aged between 6 to <18 years received a single 0.5 mL dose of 13vPnC intramuscularly on Day 1.
- Total: Total of all reporting groups
Arm/Group | 13vPnC: 6 to <18 Years | 13vPnC: 18 to <65 Years | Total
Number analyzed (Participants) | 53 | 153 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2.66) | 49.0 (10.12) | 39.6 (18.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 77 | 99
  Male | 31 | 76 | 107
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 53 | 153 | 206
  Non-Hispanic/non-Latino/not of Spanish origin | 53 | 153 | 206

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions Within 7 Days After Vaccination in Participants Aged Between 6 to <18 Years
Description: Local reactions were recorded using an electronic daily diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild (0.5 to 2.0 centimeter [cm]), moderate (greater than [>] 2.0 to 7.0 cm) and severe (>7.0 cm) for participants aged 6 to <12 years, and as mild (2.5 to 5.0 cm), moderate (>5.0 to 10.0 cm) and, severe (>10.0 cm) for participants aged 12 to <18 years. Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Day 1 up to Day 7
Population: Safety analysis set included all participants who received 1 dose of study vaccine. Here, "Number analyzed" signifies participants evaluable for each specified category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: 6 to <18 Years
Number analyzed (Participants) | 53
percentage of participants
  Redness: Any: number analyzed (Participants) | 47
  Redness: Any | 21.3 [10.7 to 35.7]
  Redness: Mild: number analyzed (Participants) | 47
  Redness: Mild | 10.6 [3.5 to 23.1]
  Redness: Moderate: number analyzed (Participants) | 47
  Redness: Moderate | 10.6 [3.5 to 23.1]
  Redness: Severe: number analyzed (Participants) | 47
  Redness: Severe | 0.0 [0.0 to 7.5]
  Swelling: Any: number analyzed (Participants) | 47
  Swelling: Any | 34.0 [20.9 to 49.3]
  Swelling: Mild: number analyzed (Participants) | 47
  Swelling: Mild | 14.9 [6.2 to 28.3]
  Swelling: Moderate: number analyzed (Participants) | 47
  Swelling: Moderate | 17.0 [7.6 to 30.8]
  Swelling: Severe: number analyzed (Participants) | 47
  Swelling: Severe | 2.1 [0.1 to 11.3]
  Pain at the injection site: Any: number analyzed (Participants) | 52
  Pain at the injection site: Any | 78.8 [65.3 to 88.9]
  Pain at the injection site: Mild: number analyzed (Participants) | 52
  Pain at the injection site: Mild | 57.7 [43.2 to 71.3]
  Pain at the injection site: Moderate: number analyzed (Participants) | 52
  Pain at the injection site: Moderate | 21.2 [11.1 to 34.7]
  Pain at the injection site: Severe: number analyzed (Participants) | 52
  Pain at the injection site: Severe | 0.0 [0.0 to 6.8]

2. Primary Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions Within 14 Days After Vaccination in Participants Aged Between 18 to <65 Years
Description: Local reactions were recorded using an electronic daily diary. Local reactions included redness, swelling and pain at injection site. Redness and swelling were graded as mild (2.5 to 5.0 cm), moderate (>5.0 to 10.0 cm) and, severe (>10.0 cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity).
Time Frame: Day 1 up to Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: 18 to <65 Years
Number analyzed (Participants) | 153
percentage of participants
  Redness: Any: number analyzed (Participants) | 135
  Redness: Any | 7.4 [3.6 to 13.2]
  Redness: Mild: number analyzed (Participants) | 135
  Redness: Mild | 5.2 [2.1 to 10.4]
  Redness: Moderate: number analyzed (Participants) | 135
  Redness: Moderate | 2.2 [0.5 to 6.4]
  Redness: Severe: number analyzed (Participants) | 135
  Redness: Severe | 0.0 [0.0 to 2.7]
  Swelling: Any: number analyzed (Participants) | 136
  Swelling: Any | 12.5 [7.5 to 19.3]
  Swelling: Mild: number analyzed (Participants) | 136
  Swelling: Mild | 5.1 [2.1 to 10.3]
  Swelling: Moderate: number analyzed (Participants) | 136
  Swelling: Moderate | 7.4 [3.6 to 13.1]
  Swelling: Severe: number analyzed (Participants) | 136
  Swelling: Severe | 0.0 [0.0 to 2.7]
  Pain at the injection site: Any: number analyzed (Participants) | 145
  Pain at the injection site: Any | 66.2 [57.9 to 73.8]
  Pain at the injection site: Mild: number analyzed (Participants) | 145
  Pain at the injection site: Mild | 53.8 [45.3 to 62.1]
  Pain at the injection site: Moderate: number analyzed (Participants) | 145
  Pain at the injection site: Moderate | 11.0 [6.4 to 17.3]
  Pain at the injection site: Severe: number analyzed (Participants) | 145
  Pain at the injection site: Severe | 1.4 [0.2 to 4.9]

3. Primary Outcome: Percentage of Participants Reporting Systemic Events and Use of Antipyretic or Pain Medication Within 7 Days After Vaccination in Participants Aged Between 6 to <18 Years
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, muscle and joint pain, and were recorded by using an e-diary. Use of antipyretic or pain medication was also collected by using an e-diary. Fever was graded as 37.5 to 38.4 degree Celsius (C), 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and >40.0 degree C. Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required intravenous hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (greater than or equals to [>=] 6 loose stools in 24 hours). Headache, fatigue, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (significant, prevented daily activity).
Time Frame: Day 1 up to Day 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: 6 to <18 Years
Number analyzed (Participants) | 53
percentage of participants
  Fever: 37.5 degree C to 38.4 degree C: number analyzed (Participants) | 48
  Fever: 37.5 degree C to 38.4 degree C | 12.5 [4.7 to 25.2]
  Fever: 38.5 degree C to 38.9 degree C: number analyzed (Participants) | 48
  Fever: 38.5 degree C to 38.9 degree C | 2.1 [0.1 to 11.1]
  Fever: 39.0 degree C to 40.0 degree C: number analyzed (Participants) | 48
  Fever: 39.0 degree C to 40.0 degree C | 0.0 [0.0 to 7.4]
  Fever: >40.0 degree C: number analyzed (Participants) | 48
  Fever: >40.0 degree C | 0.0 [0.0 to 7.4]
  Fatigue: Any: number analyzed (Participants) | 48
  Fatigue: Any | 37.5 [24.0 to 52.6]
  Fatigue: Mild: number analyzed (Participants) | 48
  Fatigue: Mild | 25.0 [13.6 to 39.6]
  Fatigue: Moderate: number analyzed (Participants) | 48
  Fatigue: Moderate | 10.4 [3.5 to 22.7]
  Fatigue: Severe: number analyzed (Participants) | 48
  Fatigue: Severe | 2.1 [0.1 to 11.1]
  Headache: Any: number analyzed (Participants) | 49
  Headache: Any | 24.5 [13.3 to 38.9]
  Headache: Mild: number analyzed (Participants) | 49
  Headache: Mild | 16.3 [7.3 to 29.7]
  Headache: Moderate: number analyzed (Participants) | 49
  Headache: Moderate | 6.1 [1.3 to 16.9]
  Headache: Severe: number analyzed (Participants) | 49
  Headache: Severe | 2.0 [0.1 to 10.9]
  Vomiting: Any: number analyzed (Participants) | 47
  Vomiting: Any | 0.0 [0.0 to 7.5]
  Vomiting: Mild: number analyzed (Participants) | 47
  Vomiting: Mild | 0.0 [0.0 to 7.5]
  Vomiting: Moderate: number analyzed (Participants) | 47
  Vomiting: Moderate | 0.0 [0.0 to 7.5]
  Vomiting: Severe: number analyzed (Participants) | 47
  Vomiting: Severe | 0.0 [0.0 to 7.5]
  Diarrhea: Any: number analyzed (Participants) | 48
  Diarrhea: Any | 8.3 [2.3 to 20.0]
  Diarrhea: Mild: number analyzed (Participants) | 48
  Diarrhea: Mild | 8.3 [2.3 to 20.0]
  Diarrhea: Moderate: number analyzed (Participants) | 48
  Diarrhea: Moderate | 0.0 [0.0 to 7.4]
  Diarrhea: Severe: number analyzed (Participants) | 48
  Diarrhea: Severe | 0.0 [0.0 to 7.4]
  Muscle pain: Any: number analyzed (Participants) | 49
  Muscle pain: Any | 30.6 [18.3 to 45.4]
  Muscle pain: Mild: number analyzed (Participants) | 49
  Muscle pain: Mild | 26.5 [14.9 to 41.1]
  Muscle pain: Moderate: number analyzed (Participants) | 49
  Muscle pain: Moderate | 4.1 [0.5 to 14.0]
  Muscle pain: Severe: number analyzed (Participants) | 49
  Muscle pain: Severe | 0.0 [0.0 to 7.3]
  Joint pain: Any: number analyzed (Participants) | 48
  Joint pain: Any | 6.3 [1.3 to 17.2]
  Joint pain: Mild: number analyzed (Participants) | 48
  Joint pain: Mild | 4.2 [0.5 to 14.3]
  Joint pain: Moderate: number analyzed (Participants) | 48
  Joint pain: Moderate | 2.1 [0.1 to 11.1]
  Joint pain: Severe: number analyzed (Participants) | 48
  Joint pain: Severe | 0.0 [0.0 to 7.4]
  Use of antipyretic or pain medication: number analyzed (Participants) | 47
  Use of antipyretic or pain medication | 6.4 [1.3 to 17.5]

4. Primary Outcome: Percentage of Participants Reporting Systemic Events and Use of Antipyretic or Pain Medication Within 14 Days After Vaccination in Participants Aged Between 18 to <65 Years
Description: Systemic events included fever, vomiting, diarrhea, headache, fatigue, muscle and joint pain, and were recorded by using an e-diary. Use of antipyretic or pain medication was also collected by using an e-diary. Fever was graded as 37.5 to 38.4 degree C, 38.5 to 38.9 degree C, 39.0 to 40.0 degree C and >40.0 degree C. Vomiting was graded as mild (1-2 times in 24 hours), moderate (>2 times in 24 hours) and severe (required intravenous hydration). Diarrhea was graded as mild (2-3 loose stools in 24 hours), moderate (4-5 loose stools in 24 hours) and severe (>=6 loose stools in 24 hours). Headache, fatigue, muscle pain and joint pain were graded as mild (no interference with activity), moderate (some interference with activity) and severe (significant, prevented daily activity).
Time Frame: Day 1 up to Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC: 18 to <65 Years
Number analyzed (Participants) | 153
percentage of participants
  Fever: 37.5 degree C to 38.4 degree C: number analyzed (Participants) | 134
  Fever: 37.5 degree C to 38.4 degree C | 6.0 [2.6 to 11.4]
  Fever: 38.5 degree C to 38.9 degree C: number analyzed (Participants) | 134
  Fever: 38.5 degree C to 38.9 degree C | 0.0 [0.0 to 2.7]
  Fever: 39.0 degree C to 40.0 degree C: number analyzed (Participants) | 134
  Fever: 39.0 degree C to 40.0 degree C | 0.0 [0.0 to 2.7]
  Fever: >40.0 degree C: number analyzed (Participants) | 134
  Fever: >40.0 degree C | 0.0 [0.0 to 2.7]
  Fatigue: Any: number analyzed (Participants) | 142
  Fatigue: Any | 33.1 [25.4 to 41.5]
  Fatigue: Mild: number analyzed (Participants) | 142
  Fatigue: Mild | 25.4 [18.4 to 33.3]
  Fatigue: Moderate: number analyzed (Participants) | 142
  Fatigue: Moderate | 7.7 [3.9 to 13.4]
  Fatigue: Severe: number analyzed (Participants) | 142
  Fatigue: Severe | 0.0 [0.0 to 2.6]
  Headache: Any: number analyzed (Participants) | 141
  Headache: Any | 23.4 [16.7 to 31.3]
  Headache: Mild: number analyzed (Participants) | 141
  Headache: Mild | 19.1 [13.0 to 26.6]
  Headache: Moderate: number analyzed (Participants) | 141
  Headache: Moderate | 4.3 [1.6 to 9.0]
  Headache: Severe: number analyzed (Participants) | 141
  Headache: Severe | 0.0 [0.0 to 2.6]
  Vomiting: Any: number analyzed (Participants) | 136
  Vomiting: Any | 1.5 [0.2 to 5.2]
  Vomiting: Mild: number analyzed (Participants) | 136
  Vomiting: Mild | 1.5 [0.2 to 5.2]
  Vomiting: Moderate: number analyzed (Participants) | 136
  Vomiting: Moderate | 0.0 [0.0 to 2.7]
  Vomiting: Severe: number analyzed (Participants) | 136
  Vomiting: Severe | 0.0 [0.0 to 2.7]
  Diarrhea: Any: number analyzed (Participants) | 141
  Diarrhea: Any | 18.4 [12.4 to 25.8]
  Diarrhea: Mild: number analyzed (Participants) | 141
  Diarrhea: Mild | 15.6 [10.0 to 22.7]
  Diarrhea: Moderate: number analyzed (Participants) | 141
  Diarrhea: Moderate | 2.1 [0.4 to 6.1]
  Diarrhea: Severe: number analyzed (Participants) | 141
  Diarrhea: Severe | 0.7 [0.0 to 3.9]
  Muscle pain: Any: number analyzed (Participants) | 139
  Muscle pain: Any | 27.3 [20.1 to 35.5]
  Muscle pain: Mild: number analyzed (Participants) | 139
  Muscle pain: Mild | 20.9 [14.4 to 28.6]
  Muscle pain: Moderate: number analyzed (Participants) | 139
  Muscle pain: Moderate | 5.8 [2.5 to 11.0]
  Muscle pain: Severe: number analyzed (Participants) | 139
  Muscle pain: Severe | 0.7 [0.0 to 3.9]
  Joint pain: Any: number analyzed (Participants) | 138
  Joint pain: Any | 13.8 [8.5 to 20.7]
  Joint pain: Mild: number analyzed (Participants) | 138
  Joint pain: Mild | 9.4 [5.1 to 15.6]
  Joint pain: Moderate: number analyzed (Participants) | 138
  Joint pain: Moderate | 3.6 [1.2 to 8.3]
  Joint pain: Severe: number analyzed (Participants) | 138
  Joint pain: Severe | 0.7 [0.0 to 4.0]
  Use of antipyretic or pain medication: number analyzed (Participants) | 134
  Use of antipyretic or pain medication | 8.2 [4.2 to 14.2]

5. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study vaccine without regard to possibility of causal relationship. An SAE is any untoward medical occurrence at any dose that results in death; is life-threatening (immediate risk of death); requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); results in congenital anomaly/birth defect.
Time Frame: signing of informed consent form (Day 1) up to Day 43
Population: Safety analysis set included all participants who received 1 dose of study vaccine.
Measure: Number; unit: percentage of participants
Groups:
- 13vPnC: All Participants: All participants aged between 6 to <65 years received a single 0.5 mL dose of 13vPnC intramuscularly on Day 1.
Arm/Group | 13vPnC: All Participants
Number analyzed (Participants) | 206
percentage of participants
  AEs | 16
  SAEs | 0

6. Secondary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) at Pre-vaccination and 1 Month After Vaccination
Description: Antibody-mediated serum OPA against each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) was measured centrally using a quantitative functional microcolony OPA (mcOPA) assay. Results were expressed as OPA titers. OPA titers were logarithmically transformed for analysis; geometric means calculated and expressed as geometric mean titers (GMTs). Two (2)-sided 95% CIs were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed based on the Student t distribution. OPA titer was expressed as reciprocal of highest serum dilution.
Time Frame: Pre-vaccination and 1 month after vaccination
Population: Evaluable immunogenicity population: eligible participants who received the study vaccine and took no prohibited vaccines, had blood drawn within 1 month after vaccination with at least 1 valid and determinate assay and had no major protocol violations. Here, "Number analyzed" signifies participants evaluable for each specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | 13vPnC: All Participants
Number analyzed (Participants) | 206
titers
  Pre-vaccination; Serotype 1: number analyzed (Participants) | 202
  Pre-vaccination; Serotype 1 | 10 [9.2 to 10.2]
  1 month after vaccination; Serotype 1: number analyzed (Participants) | 201
  1 month after vaccination; Serotype 1 | 152 [119.2 to 193.8]
  Pre-vaccination; Serotype 3: number analyzed (Participants) | 205
  Pre-vaccination; Serotype 3 | 11 [9.8 to 13.1]
  1 month after vaccination; Serotype 3: number analyzed (Participants) | 203
  1 month after vaccination; Serotype 3 | 63 [52.6 to 75.8]
  Pre-vaccination; Serotype 4: number analyzed (Participants) | 195
  Pre-vaccination; Serotype 4 | 18 [14.5 to 22.1]
  1 month after vaccination; Serotype 4: number analyzed (Participants) | 203
  1 month after vaccination; Serotype 4 | 1257 [896.0 to 1763.8]
  Pre-vaccination; Serotype 5: number analyzed (Participants) | 200
  Pre-vaccination; Serotype 5 | 16 [15.3 to 17.5]
  1 month after vaccination; Serotype 5: number analyzed (Participants) | 199
  1 month after vaccination; Serotype 5 | 185 [143.9 to 237.5]
  Pre-vaccination; Serotype 6A: number analyzed (Participants) | 171
  Pre-vaccination; Serotype 6A | 57 [44.1 to 74.9]
  1 month after vaccination; Serotype 6A: number analyzed (Participants) | 197
  1 month after vaccination; Serotype 6A | 2487 [1811.7 to 3415.0]
  Pre-vaccination; Serotype 6B: number analyzed (Participants) | 179
  Pre-vaccination; Serotype 6B | 72 [56.3 to 93.0]
  1 month after vaccination; Serotype 6B: number analyzed (Participants) | 198
  1 month after vaccination; Serotype 6B | 1845 [1405.9 to 2421.9]
  Pre-vaccination; Serotype 7F: number analyzed (Participants) | 190
  Pre-vaccination; Serotype 7F | 167 [137.0 to 203.3]
  1 month after vaccination; Serotype 7F: number analyzed (Participants) | 202
  1 month after vaccination; Serotype 7F | 2107 [1752.6 to 2532.5]
  Pre-vaccination; Serotype 9V: number analyzed (Participants) | 192
  Pre-vaccination; Serotype 9V | 204 [166.6 to 249.7]
  1 month after vaccination; Serotype 9V: number analyzed (Participants) | 199
  1 month after vaccination; Serotype 9V | 1425 [1134.4 to 1789.8]
  Pre-vaccination; Serotype 14: number analyzed (Participants) | 191
  Pre-vaccination; Serotype 14 | 129 [97.9 to 171.1]
  1 month after vaccination; Serotype 14: number analyzed (Participants) | 200
  1 month after vaccination; Serotype 14 | 1919 [1518.8 to 2424.0]
  Pre-vaccination; Serotype 18C: number analyzed (Participants) | 191
  Pre-vaccination; Serotype 18C | 61 [46.3 to 81.0]
  1 month after vaccination; Serotype 18C: number analyzed (Participants) | 199
  1 month after vaccination; Serotype 18C | 1829 [1390.8 to 2405.1]
  Pre-vaccination; Serotype 19A: number analyzed (Participants) | 202
  Pre-vaccination; Serotype 19A | 38 [29.9 to 47.8]
  1 month after vaccination; Serotype 19A: number analyzed (Participants) | 203
  1 month after vaccination; Serotype 19A | 955 [745.6 to 1223.2]
  Pre-vaccination; Serotype 19F: number analyzed (Participants) | 198
  Pre-vaccination; Serotype 19F | 42 [34.8 to 50.4]
  1 month after vaccination; Serotype 19F: number analyzed (Participants) | 197
  1 month after vaccination; Serotype 19F | 1126 [849.5 to 1493.4]
  Pre-vaccination; Serotype 23F: number analyzed (Participants) | 201
  Pre-vaccination; Serotype 23F | 14 [11.1 to 17.2]
  1 month after vaccination; Serotype 23F: number analyzed (Participants) | 202
  1 month after vaccination; Serotype 23F | 713 [506.7 to 1001.9]

7. Secondary Outcome: Geometric Mean Fold Rises (GMFRs) in Serotype-specific OPA Titers 1 Month After Vaccination
Description: OPA GMFRs were calculated along with corresponding 2-sided 95% CIs for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F. GMFRs were computed as the fold rise in titer value at 1 month after vaccination compared to baseline (pre-vaccination). The CIs for GMFRs were back transformations of a CI based on the Student t distribution for the mean difference of the log-transformed assay results before vaccination and 1 month after vaccination.
Time Frame: Pre-vaccination to 1 month after vaccination
Population: Evaluable immunogenicity set: Eligible participants received study vaccine,took no prohibited vaccine,had blood drawn in specified time frame had atleast 1 valid,determinate OPA titer/IgG concentration result for atleast 1 serotype 1 month after vaccination,no major protocol violation. Number analyzed=participant evaluable for specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC: All Participants
Number analyzed (Participants) | 206
fold rise
  Serotype 1: number analyzed (Participants) | 200
  Serotype 1 | 15.6 [12.33 to 19.82]
  Serotype 3: number analyzed (Participants) | 202
  Serotype 3 | 5.5 [4.59 to 6.54]
  Serotype 4: number analyzed (Participants) | 192
  Serotype 4 | 61.7 [42.80 to 88.99]
  Serotype 5: number analyzed (Participants) | 195
  Serotype 5 | 11.2 [8.69 to 14.34]
  Serotype 6A: number analyzed (Participants) | 167
  Serotype 6A | 34.7 [24.39 to 49.44]
  Serotype 6B: number analyzed (Participants) | 174
  Serotype 6B | 21.9 [15.71 to 30.51]
  Serotype 7F: number analyzed (Participants) | 188
  Serotype 7F | 12.1 [9.84 to 14.76]
  Serotype 9V: number analyzed (Participants) | 188
  Serotype 9V | 6.8 [5.36 to 8.62]
  Serotype 14: number analyzed (Participants) | 186
  Serotype 14 | 13.2 [9.63 to 18.04]
  Serotype 18C: number analyzed (Participants) | 186
  Serotype 18C | 26.7 [19.39 to 36.86]
  Serotype 19A: number analyzed (Participants) | 199
  Serotype 19A | 24.9 [19.05 to 32.66]
  Serotype 19F: number analyzed (Participants) | 192
  Serotype 19F | 26.6 [19.89 to 35.63]
  Serotype 23F: number analyzed (Participants) | 200
  Serotype 23F | 50.4 [35.70 to 71.16]

8. Secondary Outcome: Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentrations (GMCs) at Pre-vaccination and 1 Month After Vaccination
Description: Pneumococcal IgG antibody against each of the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) was measured centrally using direct binding Luminex assay. Results were expressed as IgG concentrations. IgG concentrations were logarithmically transformed for analysis; geometric means calculated and expressed as GMCs. Two (2)-sided 95% CIs were constructed by back transformation of the CI for the mean of the logarithmically transformed assay results computed based on the Student t distribution.
Time Frame: Pre-vaccination and 1 month after vaccination
Population: Evaluable immunogenicity set: Eligible participants received study vaccine, took no prohibited vaccine, had blood drawn in specified time frame had atleast 1 valid, determinate OPA titer/IgG concentration result for atleast 1 serotype 1 month after vaccination, no major protocol violation.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC: All Participants
Number analyzed (Participants) | 206
microgram per milliliter (mcg/mL)
  Pre-vaccination; Serotype 1 | 0.132 [0.109 to 0.161]
  1 month after vaccination; Serotype 1 | 4.427 [3.423 to 5.726]
  Pre-vaccination; Serotype 3 | 0.115 [0.094 to 0.141]
  1 month after vaccination; Serotype 3 | 0.531 [0.437 to 0.646]
  Pre-vaccination; Serotype 4 | 0.055 [0.045 to 0.068]
  1 month after vaccination; Serotype 4 | 1.826 [1.387 to 2.404]
  Pre-vaccination; Serotype 5 | 0.058 [0.046 to 0.075]
  1 month after vaccination; Serotype 5 | 2.779 [1.972 to 3.915]
  Pre-vaccination; Serotype 6A | 0.173 [0.133 to 0.224]
  1 month after vaccination; Serotype 6A | 4.070 [2.915 to 5.684]
  Pre-vaccination; Serotype 6B | 0.105 [0.080 to 0.138]
  1 month after vaccination; Serotype 6B | 2.354 [1.631 to 3.396]
  Pre-vaccination; Serotype 7F | 0.117 [0.092 to 0.150]
  1 month after vaccination; Serotype 7F | 4.670 [3.629 to 6.010]
  Pre-vaccination; Serotype 9V | 0.067 [0.054 to 0.082]
  1 month after vaccination; Serotype 9V | 1.483 [1.131 to 1.944]
  Pre-vaccination; Serotype 14 | 0.335 [0.252 to 0.447]
  1 month after vaccination; Serotype 14 | 7.769 [5.844 to 10.328]
  Pre-vaccination; Serotype 18C | 0.168 [0.131 to 0.216]
  1 month after vaccination; Serotype 18C | 5.187 [4.026 to 6.682]
  Pre-vaccination; Serotype 19A | 0.496 [0.391 to 0.629]
  1 month after vaccination; Serotype 19A | 7.616 [5.786 to 10.026]
  Pre-vaccination; Serotype 19F | 0.217 [0.171 to 0.275]
  1 month after vaccination; Serotype 19F | 4.315 [3.241 to 5.744]
  Pre-vaccination; Serotype 23F | 0.181 [0.143 to 0.228]
  1 month after vaccination; Serotype 23F | 6.283 [4.524 to 8.727]

9. Secondary Outcome: GMFRs in Serotype-specific IgG From Before Vaccination to 1 Month After Vaccination
Description: IgG GMFRs were calculated along with corresponding 2-sided 95% CIs for pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F. GMFRs were computed as the fold rise in concentrations at 1 month after vaccination compared to baseline (pre-vaccination). The CIs for GMFRs were back transformations of a CI based on the Student t distribution for the mean difference of the log-transformed assay results before vaccination and 1 month after vaccination.
Time Frame: Pre- vaccination to 1 month after vaccination
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC: All Participants
Number analyzed (Participants) | 206
fold rise
  Serotype 1 | 33.445 [26.374 to 42.413]
  Serotype 3 | 4.605 [3.839 to 5.524]
  Serotype 4 | 32.960 [25.331 to 42.886]
  Serotype 5 | 47.565 [36.867 to 61.368]
  Serotype 6A | 23.587 [18.010 to 30.890]
  Serotype 6B | 22.421 [17.045 to 29.493]
  Serotype 7F | 39.843 [31.473 to 50.438]
  Serotype 9V | 22.232 [17.426 to 28.362]
  Serotype 14 | 23.161 [17.179 to 31.227]
  Serotype 18C | 30.833 [24.008 to 39.597]
  Serotype 19A | 15.354 [12.116 to 19.459]
  Serotype 19F | 19.892 [15.552 to 25.443]
  Serotype 23F | 34.809 [26.436 to 45.833]

ADVERSE EVENTS:
Time Frame: signing of informed consent form (Day 1) up to Day 43
Arm/Group | 13vPnC: 6 to <18 Years | 13vPnC: 18 to <65 Years | 13vPnC: All Participants
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/153 | 0/206
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/153 | 0/206
Other Adverse Events (participants affected / at risk) | 49/53 | 121/153 | 170/206
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC: 6 to <18 Years (N=53) | 13vPnC: 18 to <65 Years (N=153) | 13vPnC: All Participants (N=206)
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 4/48 | 26/141 | 30/189 — Number of participants at risk = number of participants evaluable for the adverse event.
Vomiting (Gastrointestinal disorders) | 0/47 | 2/136 | 2/183 — Number of participants at risk = number of participants evaluable for the adverse event.
Fatigue (General disorders) | 18/48 | 47/142 | 65/190 — Number of participants at risk = number of participants evaluable for the adverse event.
Redness (General disorders) | 10/47 | 10/135 | 20/182 — Number of participants at risk = number of participants evaluable for the adverse event.
Injection site erythema (General disorders) | 1 | 0 | 1
Pain at the injection site (General disorders) | 41/52 | 96/145 | 137/197 — Number of participants at risk = number of participants evaluable for the adverse event.
Injection site pain (General disorders) | 1 | 2 | 3
Injection site swelling (General disorders) | 16/47 | 17/136 | 33/183 — Number of participants at risk = number of participants evaluable for the adverse event.
Pyrexia (General disorders) | 7/48 | 8/134 | 15/182 — Number of participants at risk = number of participants evaluable for the adverse event.
Bronchitis (Infections and infestations) | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 8 | 9
Pharyngitis (Infections and infestations) | 3 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/48 | 19/138 | 22/186 — Number of participants at risk = number of participants evaluable for the adverse event.
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 15/49 | 38/139 | 53/188 — Number of participants at risk = number of participants evaluable for the adverse event.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 12/49 | 33/141 | 45/190 — Number of participants at risk = number of participants evaluable for the adverse event.
Middle insomnia (Psychiatric disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03571607/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT03571607/SAP_001.pdf